CLINICAL TRIAL: NCT06885632
Title: The Effectiveness of Probiotic Gummies in Relieving Allergic Rhinitis in Children and Their Regulatory Effect on the Gut Microbiota and Metabolic Profile
Brief Title: Effectiveness of Probiotic Gummies in Relieving Allergic Rhinitis in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK20250314
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Children With Allergic Rhinitis
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Probiotic pectin gummies(500 million CFU)/2 pellets/day BC99
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): No probiotic pectin gummies/2 pellets/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of this study lasts 56 days and each patient will have 3 visits (week0, week4, week8).
  Arms: Probiotic group
Dietary Supplement: Placebo — The experimental phase of this study lasts 56 days and each patient will have 3 visits (week0, week4, week8).
  Arms: Placebo group

SUMMARY:
To evaluate the effect of probiotic gummies on serum metabolite levels, clinical efficacy, and regulation of gut microbiota in children with allergic rhinitis compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary, written, signed informed consent to participate in this study;
2. be able to complete the study in accordance with the requirements of the test protocol;
3. Age 4-14 years old;
4. Meet the diagnostic criteria for allergic rhinitis established in the Guidelines for the Diagnosis and Treatment of Allergic Rhinitis in Children (2022 Revised Edition);
5. Symptoms: 2 or more symptoms: sneezing, watery discharge, nasal itching and nasal congestion and other symptoms last or accumulate for more than 1 hour per day, and may be accompanied by eye symptoms such as itching, watery eyes and red eyes;
6. Signs: pale and edema of the nasal mucosa, which may be accompanied by watery discharge;

Exclusion Criteria:

1. Drugs that affect the intestinal flora (including antimicrobial drugs, microecological preparations, intestinal mucosal protectors, Chinese patent medicines, etc.) have been used continuously for more than 1 week within 1 month before screening;
2. Patients with pulmonary tuberculosis;
3. Combined with allergic asthma;
4. Those with nasal polyps or severe nasal septum deviation;
5. Patients with severe systemic diseases or malignant tumors;
6. Those with congenital genetic diseases and congenital immunodeficiency diseases;
7. Those who regularly use probiotics or prebiotics within 6 months before the screening period;
8. Those with severe digestive tract diseases (including severe diarrhea, inflammatory bowel disease, etc.);
9. Patients with metabolic syndrome (including obesity, dyslipidemia, hypertension, diabetes, etc.);
10. Patients with sinusitis, otitis media, or respiratory tract infection;
11. Those who are allergic to the probiotic-related ingredients used in this trial;
12. Those who stop taking the test sample or add other drugs in the middle of the test, and the efficacy cannot be judged or the data is incomplete;
13. Those who take items with similar functions to the test in a short period of time, which affects the judgment of the results;
14. Subjects who are unable to participate in the test due to their own reasons;
15. Subjects who are judged by other investigators to be insuitable to participate.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Changes in the structure of fecal microbiota before and after the intervention. | Week 0 and Week 8
  Analyzed by 16S rRNA sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- The School of Food and Bioengineering, Henan University of Science and Technolog, Luoyang, Henan, China